CLINICAL TRIAL: NCT03114748
Title: Monitoring électroencéphalographique Chez Les Patients traités Par Stimulation cérébrale Profonde
Brief Title: Electroencephalographic Monitoring in Patients Treated by Deep Brain Stimulation
Acronym: EEG-DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012-A00490-43
Record Dates: First submitted 2017-02-08; First posted 2017-04-14 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-07

CONDITIONS: Motor Disorders; Psychiatric Disorder
Keywords: deep brain stimulation; EEG
MeSH Terms: conditions — Motor Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EEG (Experimental): 2 scalp electroencephalographic (EEG) recording will be acquired in ON and OFF DBS conditions
  Interventions: Other: EEG
- DBS ON and OFF (Experimental): DBS is turned ON and OFF in the 2 EEG sections
  Interventions: Other: DBS switched OFF and ON

INTERVENTIONS:
Other: EEG
  Arms: EEG
Other: DBS switched OFF and ON
  Arms: DBS ON and OFF

SUMMARY:
This protocol aims to develop the use of behavioral and electroencephalographic measures during cognitive tasks in patients treated with deep brain stimulation during the stimulation parameters adjustments. The main clinical goal of this protocol is to find behavioral and or electroencephalographic markers to evaluates the right targeting of stimulation electrodes. On the more fundamental point of view, the study of those data can be used to understand better the action mechanisms of deep brain stimulation.

DETAILED DESCRIPTION:
This protocol aims to understand how brain regions are modulated by deep brain stimulation using scalp electroencephalographic recordings. This protocol covers many pathologies which are thought to relate to different brain networks impairements and are therefore complementary in the understanding of cortical activation and modulation of this activation by deep brain stimulation. These diseases are motor (parkinson..) and psychiatric (obsessive compulsive disorders, treatment resistant depression..). To activate brain networks of interest, either implicating brain regions dysfunctional in the diseases or brain regions stimulated by the electrode, the investigators can use cognitive task which are know to involve those networks, for instance motor task for motor diseases as clicking with a computer mouse when presented with a specific type of stimulus on the screen. EEG recordings can then be processed to retrieve cortical activation and modulation of this activation with stimulation (using an ON DBS OFF DBS procedure) during task processing. These data are also very precious to study brain dynamic networks and their modulation by DBS. After analysis of these results, this protocol aims to be used in order to refine targeting, for instance when correlating cortical modulation with DBS and clinical improvement with electrode positions.

ELIGIBILITY:
Inclusion Criteria:

* patient treated with DBS
* study inclusion written agreement by the patient or his legal representant
* intellectual capacities compatible with cognitive task and EEG recordings
* French native speaker and capacity to understand the study processes and particularly to fill in the auto questionaires
* patients abled to give an enlighted agreement
* patients who have an health insurance coverage

Exclusion Criteria:

* people who fill in the articles L1121-5 to L1121-8 or the Public Health Code
* patients who don't stand the transient interruption of stimulation
* severe concomitant disease
* disease which impose a treatment which modulates vigilance
* cognitive alteration (Mattis<130)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2019-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
EEG recordings from 96 scalp electrodes | around 15 minutes for each condition
  high resolution voltage signal from the patients scalp

CONTACTS AND LOCATIONS:
Overall Officials: Stephan CHABARDES, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No